CLINICAL TRIAL: NCT04267874
Title: The BE WELL Study: Black Raspberry Beverage Working to Prevent Lung Cancer
Brief Title: Black Raspberry Nectar for the Prevention of Lung Cancer, BE WELL Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Daniel Spakowicz, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: OSU-19007; NCI-2020-00418 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Lung Carcinoma; Tobacco-Related Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (BRB nectar, placebo, biospecimen collection) (Experimental): Patients receive BRB nectar PO BID for weeks 0-4 and then receive placebo PO BID for weeks 6-10 in the absence of unacceptable toxicity. Patients also undergo collection of nasal swabs, blood, urine, and stool samples at weeks 0, 4, 6, and 10.
  Interventions: Procedure: Biospecimen Collection; Dietary Supplement: Nutritional Supplementation; Drug: Placebo Administration; Other: Questionnaire Administration
- Arm II (placebo, BRB nectar, biospecimen collection) (Experimental): Patients receive placebo PO BID for weeks 0-4 and then receive BRB nectar PO BID for weeks 6-10 in the absence of unacceptable toxicity. Patients also undergo collection of nasal swabs, blood, urine, and stool samples at weeks 0, 4, 6, and 10.
  Interventions: Procedure: Biospecimen Collection; Dietary Supplement: Nutritional Supplementation; Drug: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of nasal swabs, blood, urine, and stool
Dietary Supplement: Nutritional Supplementation — Given black raspberry nectar PO
  Other Names: supplementation
Drug: Placebo Administration — Given PO
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well black raspberry nectar works in changing the gut microbiome and in reducing inflammatory processes that may lead to lung cancer. Studying the effects of black raspberry beverage on inflammation may help doctors find strategies to reduce the risk of developing lung cancer.

DETAILED DESCRIPTION:
PRIMARY FEASIBILITY OBJECTIVE:

I. To evaluate the feasibility of establishing a diet intervention trial with longitudinal microbiome collection in Ohio State University Comprehensive Cancer Center (OSUCCC) Lung Cancer Screening Clinic (OSUCCC-LCSC).

PRIMARY SCIENTIFIC OBJECTIVE:

I. To determine the impact of the black raspberry (BRB) nectar intervention on the microbiome and inflammatory biomarkers.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive BRB nectar orally (PO) twice daily (BID) for weeks 0-4 and then receive placebo PO BID for weeks 6-10 in the absence of unacceptable toxicity. Patients also undergo collection of nasal swabs, blood, urine, and stool samples at weeks 0, 4, 6, and 10.

ARM II: Patients receive placebo PO BID for weeks 0-4 and then receive BRB nectar PO BID for weeks 6-10 in the absence of unacceptable toxicity. Patients also undergo collection of nasal swabs, blood, urine, and stool samples at weeks 0, 4, 6, and 10.

ELIGIBILITY:
Inclusion Criteria:

* Have a 30 pack-year smoking history
* Be either a current smoker or a former smoker that quit in the last 15 years. Any individual who is currently smoking and has smoked more than 100 cigarettes in their lifetime will be identified as a current smoker
* Agree to consume a standardized vitamin / mineral supplement and avoid other nutritional, dietary or alternative medications / supplements / probiotics for the duration of the study
* Agree to follow a berry-free / controlled phenolic diet and to document consumption of polyphenolic foods each day of the study using a simple daily form

Exclusion Criteria:

* Person has an allergy to any berries, pectin, or food colorants apples,as well as kiwi fruit, strawberries, soy sauce, pine nuts, almonds, cherries, peaches, blackberries, pears
* Person states that they are not a:

  * Current smoker: active cigarette smoker who has smoked more than 30 pack-years in the last 15 years OR
  * Former smoker: not a current smoker active cigarette smoker who has smoked more than 30 pack years in the last 15 years
* Person is unwilling to follow a berry-free/controlled polyphenol diet while on study
* Person has history of metabolic disorders (diabetes, hyper/hypo-thyroidism, etc.); digestive illness which may result in nutrient malabsorption (Crohn's disease, Celiac, renal/hepatic insufficiency, short bowel, etc.); disorders that affect connective tissues; or blood clotting disorders
* Person has allergy or food intolerance to ingredients in study products (black raspberries or other berries)
* Person is on a regimen of any of the following medications:

  * Immunosuppressants, bisphosphonates, or steroids.
  * Anticoagulants (warfarin, apixaban, dabigatran, and rivaroxaban)
  * Probiotics
* Person is undergoing treatment for cancer in any form
* Person is currently pregnant or nursing or plans to become pregnant during this study
* Person plans to enter smoking cessation or change their smoking status during the course of the study

Ages: 55 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-06-13 (Actual)

PRIMARY OUTCOMES:
Recruitment rates | Up to 3 years
  Recruitment rates will be defined as the proportion of screened accrued relative to those approached. Successful recruitment rates will be defined as >= 10% of participants approached agree to participate.
Study adherence | Up to 3 years
  Study adherence will be defined as the percent of the biospecimens collected at the end of the study period, with a compliance goal of 60%. Will track the monthly collection of data and document reasons for missing any scheduled collection dates. The proportions of missing information at each time point will be calculated. Descriptive statistics will examine the distribution of all patient and treatment characteristics, overall and by patient and disease characteristics.
Inflammatory markers found in nasal brushings | Up to 3 years
  Evaluated by ribonucleic acid sequencing.
Changes in stool microbe relative abundances | Up to 3 years
  Evaluated by metagenomic whole sequencing.
Biologic responses to the black raspberry (BRB) nectar | Up to 3 years
  Samples of urine, stool. and blood will be analyzed for BRB phytochemicals (ellagitannins, ellagic acid, quercetin glycosides, anthocyanins) and their metabolites (urolithins, quercetin glucuronides/sulfates, methylated anthocyanins).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Spakowicz, PhD, MS, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Informed Consent Form (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT04267874/ICF_000.pdf